CLINICAL TRIAL: NCT05008679
Title: The Effects of Neuraminidase Inhibitor Oseltamivir in Patients With Chronic Heart Failure: an Open Label, Randomized, Blank-controlled Study.
Brief Title: The Effects of Neuraminidase Inhibitor Oseltamivir in Patients With Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-HF-NI
Record Dates: First submitted 2021-08-14; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
Keywords: heart failure; Neuraminidase inhibitor; oseltamivir; Neu5Ac; NTproBNP
MeSH Terms: conditions — Heart Failure | interventions — Oseltamivir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): patients with heart failure to receive standard HF therapy
- Oseltamivir (Experimental): patients with heart failure to receive oseltamivir (at a dose of 75 mg twice daily) for 1 month in addition to standard HF therapy
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — at a dose of 75 mg twice daily
  Other Names: Neuraminidase Inhibitor
  Arms: Oseltamivir

SUMMARY:
Heart failure (HF) is a complex syndrome with increasing incidence and high rates of mortality and hospitalization. Although inhibitors of angiotensin converting enzyme (ACE), β-blockers and aldosterone-receptor blockers have improved the treatment of heart failure, mortality of HF remains unacceptably high.

Recently, we identified a key metabolite N-acetylneuraminic acid (Neu5Ac) increased in the plasma of patients with heart failure. Also, elevated plasma Neu5Ac, independent of other traditional risk factors, is associated with poor prognosis in patients with HF in long-term follow up. Neu5Ac levels, the most common sialic acid in mammals, generated from sialylated glycoconjugates by neuraminidase. Neu5Ac and its regulatory enzyme neuraminidase play a key role in heart failure. We found neuraminidase inhibitor could reduce Neu5Ac levels and improve heart failure in mice model, providing opportunity for a novel therapeutic strategy in HF. Neuraminidase inhibitor oseltamivir is also an old anti-influenza drug. Using oseltamivir may be a new therapeutic strategy in heart failure.

Based on above information, we designed the randomized, open-label, blank-controlled study in patients with chronic HF to receive either oseltamivir or placebo, in addition to standard HF therapy to Identify the effect of oseltamivir on serum Neu5Ac level in patients with heart failure and assess the clinic outcomes of level in patients with heart failure using oseltamivir.

ELIGIBILITY:
Inclusion Criteria:

1. 18 of age or older, regardless of gender;
2. Patients with NYHA II-IV, LVEF less than 40%;
3. Levels of NT-proBNP more than 450 pg/ml
4. Willing to participate in this study and sign an informed consent, and receive follow-up contact for at least 6 months.

Exclusion Criteria:

1. Onset of acute myocardial infarction within the last 1 month;
2. Had cardiac surgery or onset of cerebrovascular accident within the last 6 months;
3. Plan to have cardiac transplantation or CRT, or already having CRT therapy;
4. Females with pregnancy or plan to have pregnancy;
5. Have participate in any other clinical trial within the last 3 months;
6. Severe neurological disorders (Alzheimer's disease, progressive stage of Parkinson's syndrome), disabilities of lower limbs or deaf-mute;
7. had a history of tumour, or precancerous lesions confirmed by pathological tests (ductal carcinoma in situ, cervical dysplasia, etc.);
8. had malignant tumours (by physical examinations, X-ray, type-B ultrasonic imaging or other methods), or had hyperplastic glands or adenoma which possess endocrine activity and affect cardiac or endocrine functions (pheochromocytoma, goitre, etc.);
9. The subjects who refuse to comply with the items of the research protocol;
10. The subjects who are not available to fulfil the follow-up plan (due to project management or other reasons), according to the judgement of researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-02-25 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP | 1 month
  Reduction of NT-proBNP level at 1 month treatment of Oseltamivir

SECONDARY OUTCOMES:
EF (ejection fraction) | 1month, 6 months
  Cardiac systolic function assessed by ejection fraction using echocardiography
NYHA Classification | 1month, 6 months
  NYHA Classification after treatment of Oseltamivir
Quality of life assessment | 1month, 6 months
  Minnesota Heart Failure Quality of life assessment after treatment of Oseltamivir
6-minute walk test | 1month, 6 months
  6-minute walk test after treatment of Oseltamivir

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China